CLINICAL TRIAL: NCT04230642
Title: Multicenter Study to Evaluate the Safety and Performance of the Quantum Surgical Robotic Device for Image-guided Percutaneous Needle Placement
Brief Title: Multicenter Study to Evaluate a New Robotic Device for Image-guided Percutaneous Needle Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QS-IS-G-H-1901
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hepatic Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic device (Experimental): Needle placement to the tumor, one time, the day of the ablation procedure
  Interventions: Device: The Quantum Surgical device

INTERVENTIONS:
Device: The Quantum Surgical device — Robotic platform for needle placement

SUMMARY:
This study evaluates the safety and performance of a new robotic device in the treatment of hepatic thermoablation in adults. The new robotic device will be used in all patients.

DETAILED DESCRIPTION:
The device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of needle, as well as in verification of needle position during CT guided percutaneous ablation procedures.

After validation of the correct positioning of the needle, the tumor ablation procedure is conducted with a device routinely used by the investigator. The Acquisition of a post-interventional CT-guided image is realized to evaluate adverse events occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old,
* Patient for whom an ablation procedure under CT guidance in liver organ has been prescribed and consensually agreed by a multidisciplinary team of radiologists, surgeons and clinicians,
* Patient not taking platelet antiaggregant or having stopped taking it for 5 days and not taking anticoagulant (thrombocytes ≥ 50 000/mm3, TP > 50%),
* Patient who agrees to participate in the evaluation and who has signed the inform consent,
* Patient covered by social security system.

Exclusion Criteria:

* Patient unable to undergo general anesthesia,
* Patient unable to tolerate CT contrast agent
* Patient already participating in another clinical study
* Pregnant or breast-feeding woman.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety related to the procedure | During the procedure
  Number of Adverse Event(s) that are considered to be major and are attributable to the needle insertion phase of the procedure
Evaluation of the feasibility of the Quantum Surgical device: Number of targets reached | During the procedure
  Number of targets reached; the target is considered to have been reached when the needle is positioned accurately enough to allow the next step of the procedure to be carried out

SECONDARY OUTCOMES:
Evaluation of the accuracy of the device | Through study completion, an average of 1 month
  Assessment of the needle placement accuracy (distance from the needle tip to the target)
Evaluation of the needle readjustments of the device | During the procedure
  Assessment of the number of needle readjustments to reach the target
Evaluation of the safety not related to the procedure | Through study completion, an average of 1 month
  All Adverse Event(s) except those considered major and are attributable to the needle insertion phase of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Boris Guiu, MD, Principal Investigator — Head of radiology department
Locations (2):
- France (2):
  - Chu Montpellier, Montpellier
  - Gustave Roussy Institut, Villejuif

IPD SHARING:
Plan to Share IPD: No